CLINICAL TRIAL: NCT04842136
Title: Comparison of Factors Affecting Patients With a Myofascial Temporomandibular Disorder With and Without Sleep Bruxism
Brief Title: Factors Affecting Patients With Myofascial Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, PT, PhD, Hasan Kalyoncu University
Other Study IDs: 2020/026
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Myofascial Temporomandibular Disorder; Bruxism, Sleep; Sleep Disturbance; Jaw Spasm; Headache
Keywords: Temporomandibular Disorders; Sleep bruxism; Neck Disability; Sleep; Headache
MeSH Terms: conditions — Sleep Bruxism; Parasomnias; Tetanus; Headache; Temporomandibular Joint Disorders | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myofascial Temporomandibular Disorder (TMD) with Sleep Bruxism (SB): Patients with Myofascial TMD and with sleep bruxism with the diagnosis of regular or frequent teeth grinding sounds during the sleep, and one or more following clinical signs, such as jaw muscle pain or fatigue on waking up in the morning, temporal headache, hypertrophy of the masseter muscle, abnormal tooth wear, and/or jaw locking were included in the group.
  Interventions: Other: Scales and indexes
- Myofascial Temporomandibular Disorder (TMD) without Sleep Bruxism (SB): Patients with Myofascial TMD without sleep bruxism were included in the group.
  Interventions: Other: Scales and indexes

INTERVENTIONS:
Other: Scales and indexes — Patients with TMD regardless of diagnosis with sleep bruxism were assessed with the Jaw Function Limitations Scale (JFLS), Neck Disability Index (NDI), Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), and Headache Impact Test-6 (HIT-6) scales.

SUMMARY:
The aim of the study was to assess and compare the relationship between jaw function, neck disability, sleep quality, fatigue, and headache in patients with myofascial Temporomandibular Disorder (TMD) with Sleep Bruxism (SB) and without (non-SB).

DETAILED DESCRIPTION:
The study was conducted on TMD patients who were willing to participate in the study between January and December 2020.

The case-control study included patients diagnosed with myofascial TMD by dental practitioners at regional hospitals referred for physiotherapy. Total of 200 myofascial TMD patients, comprising 91 identified as SB and 109 as non-SB were included in the study.

The Jaw Function Limitations Scale (JFLS), Neck Disability Index (NDI), Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), and Headache Impact Test-6 (HIT-6) scales and indexes were used for both groups.

The effect of Sleep Bruxism (SB) on jaw function, neck problems, sleep quality, fatigue, and tension headache were evaluated.

The interactions of these factors and the importance of taking SB into consideration when evaluating and treating patients with TMD were examined.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of myofascial TMD according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
* pain for more than 6 months
* no therapeutic interventions reported for TMD or the neck in the last 6 months
* intellectual capacity to provide informed consent

Exclusion Criteria:

* not meeting the DC/TMD criteria
* diagnosis of psychiatric disease
* history of surgery related to the cervical region and/or TMJ
* cervical and/or TMJ malignancy
* trauma history
* proven specific pathologies such as fracture, or rheumatoid disease
* history of facial paralysis
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a chief complaint of pain and functional limitation at the temporomandibular region were assessed by dentists at regional hospitals. Those who were diagnosed with myofascial TMD according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) participated in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  The severity of pain in muscles was measured in centimeters using a 0-10 Visual Analogue Scales (VAS). The scale ranges from 0 = "no pain at all" to 10 = "intolerable pain"
Jaw Functional Limitation Scale | Baseline
  The Jaw Functional Limitation Scale-20 was used to assess jaw function in the masticatory system. The scale consists of a total of 20 items with three constructs. Each item is scored from 0-10, with 0 indicating no restriction and 10, severe restriction. A total of ≥5 indicates jaw function limitation.
Neck Disability Index | Baseline
  Neck problems were assessed with Neck Disability Index (NDI). It is a scale of 10 sections with total points ranging from 0-50. Higher scores indicate severe pain, and a score of ≥5 indicates a neck disorder.
Pittsburgh Sleep Quality Index | Baseline
  The sleep quality was evaluated using the Pittsburgh Sleep Quality Index (PSQI). The scale comprises a total of 24 items in 7 sub-scales. The total points of the 19 items that score from 0-21, with a total of ≥5 indicating poor sleep quality.
Fatigue Severity Scale | Baseline
  The effect of fatigue on functional and behavioral aspects was evaluated by the Fatigue Severity Scale (FSS). The total score is calculated as the average of the 9 item scores -the lower the total score, the lower the fatigue level. A cut-off value of ≥4 has been defined for fatigue
Headache Impact Test | Baseline
  The Headache Impact Test-6 (HİT-6) was used to assess the headache. The 6 items scale evaluating the frequency, the degree of restriction to daily life and social life, and changes in the mood because of headache. The total score 50-59 reflects important impact, and scores ≥60 indicate severe impact.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, Study Director — Hasan Kalyoncu University
Locations (2):
- Turkey (Türkiye) (2):
  - Abdulkadir Konukoglu Healthy Life Center, Gaziantep
  - Umut Rehabilitation Center, Sanliurfa

IPD SHARING:
Plan to Share IPD: No